CLINICAL TRIAL: NCT00438841
Title: A Phase II Trial With VELCADE® (PS-341), Cytoxan (Cyclophosphamide), Dexamethasone and Thalomid® (VEL-CTD) in Previously Untreated Multiple Myeloma Patients
Brief Title: Bortezomib, Cyclophosphamide, Dexamethasone, and Thalidomide in Treating Patients With Newly Diagnosed, Previously Untreated Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Phyllis Potts, Aptium Oncology
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000536219; FHCRC-2123.00
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Cyclophosphamide; Dexamethasone; Thalidomide

INTERVENTIONS:
Drug: bortezomib
Drug: cyclophosphamide
Drug: dexamethasone
Drug: thalidomide

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cyclophosphamide and dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Thalidomide may stop the growth of cancer cells by blocking blood flow to the cancer. Giving bortezomib together with cyclophosphamide, dexamethasone, and thalidomide may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with cyclophosphamide, dexamethasone, and thalidomide works in treating patients with newly diagnosed, previously untreated multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with newly diagnosed, previously untreated multiple myeloma treated with bortezomib, cyclophosphamide, dexamethasone, and thalidomide.

Secondary

* Determine the safety and tolerability of this regimen in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive bortezomib IV on days 1, 4, 8, and 11; cyclophosphamide IV on days 1 and 8 of courses 1-3; oral thalidomide once daily on days 1-21 beginning in course 4; and dexamethasone IV or orally once daily on days 1, 2, 4, 5, 8, 9, 11, and 12. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma meeting 1 of the following criteria:

  * Monoclonal immunoglobulin spike on serum electrophoresis (IgG > 3.5 g/dL or IgA > 2.0 g/dL) and kappa or lambda light chain excretion > 1 g/day by 24-hour urine protein electrophoresis AND meets any of the following criteria:

    * Bone marrow plasmacytosis (10-30% plasma cells)
    * Lytic bone lesions
  * Monoclonal immunoglobulin of lesser magnitude present and bone marrow plasmacytosis (10-30% plasma cells) AND meets any of the following criteria:

    * Lytic bone lesions
    * IgM < 50 mg/dL, IgA < 100 mg/dL, or IgG < 600 mg/dL
  * Bone marrow plasmacytosis (> 30% plasma cells) or plasmacytoma on tissue biopsy AND meets any of the following criteria:

    * Monoclonal immunoglobulin of lesser magnitude present
    * Lytic bone lesions
    * IgM < 50 mg/dL, IgA < 100 mg/dL, or IgG < 600 mg/dL
  * FreeLite testing abnormal and kappa:lambda light chain ratio abnormal
* Symptomatic disease requiring treatment

  * Documented related organ or tissue involvement, if present
* Measurable disease, defined as 1 of the following:

  * Monoclonal immunoglobulin spike on serum electrophoresis ≥ 1 g/dL and/or urine monoclonal immunoglobulin spike ≥ 200 mg/day
  * Abnormal FreeLite testing (for nonsecretors)
  * Patients with nonsecretory disease must meet either of the following criteria for measurability:

    * Has measurable protein by FreeLite testing
    * Untreated soft tissue plasmacytoma and/or evaluable disease in bone marrow
* Newly diagnosed, previously untreated disease
* No POEMS syndrome (i.e., plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein [M-protein], and skin changes)
* No plasma cell leukemia

PATIENT CHARACTERISTICS:

* Karnofsky performance status 50-100%
* Platelet count ≥ 100,000/mm³ (≥ 50,000/mm³ if bone marrow is extensively infiltrated)

  * Extensive infiltration is defined as > 50% myeloma cells or plasma cells
* Hemoglobin ≥ 8.5 g/dL
* Absolute neutrophil count ≥ 1,500/mm³
* AST and ALT ≤ 2 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN (unless clearly related to the disease)
* Creatinine clearance ≥ 20 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception ≥ 4 weeks prior to beginning treatment, during, and for ≥ 4 weeks after completion of study treatment
* No impaired kidney function requiring dialysis
* No uncontrolled infection
* No HIV positivity
* No known active hepatitis B or C
* No cardiovascular disease including, but not limited to, any of the following:

  * Myocardial infarction within the past 6 months
  * New York Heart Association class II-IV heart failure
  * Uncontrolled angina
  * Severe uncontrolled ventricular arrhythmias
  * Clinically significant pericardial disease
  * Acute ischemic or active conduction system abnormalities by EKG
* No history of allergic reactions to compounds containing mannitol, bortezomib, or cyclophosphamide
* No second malignancy requiring concurrent treatment
* No other serious medical or psychiatric illness that would preclude study compliance
* No peripheral neuropathy ≥ grade 1

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, immunotherapy, vaccine therapy, therapeutic doses of steroids, or other agents for the treatment of active myeloma

  * Drugs given to prevent onset of myeloma allowed
  * Bisphosphonates for hypercalcemia or short course corticosteroids for hypercalcemia or cord compromise allowed
* Prior local radiotherapy with or without a brief exposure to steroids allowed
* More than 4 weeks since prior and no concurrent radiotherapy

  * Spot radiotherapy to ≤ 3 vertebrae allowed
* No concurrent steroids at > 10 mg of prednisone daily (or the equivalent) for other medical conditions (e.g., asthma, systemic lupus erythematosus, or rheumatoid arthritis)
* No other concurrent chemotherapy or investigational agents
* Concurrent daily acetylsalicylic acid required during course 4-6 of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: William I. Bensinger, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (10):
- United States (10):
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Sutter Cancer Center, Sacramento, California
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - St. Vincent's Comprehensive Cancer Center - Manhattan, New York, New York
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - Lone Star Oncology - Austin, Austin, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington